# CMSL Ambulatory Sensitive Condition Nudge (pending)

Study Protocol with Statistical Analysis Plan

January 24, 2025

#### Study Protocol

### **Background and Objective**

The project aims to evaluate a nurse-led intervention to reduce inappropriate emergency department (ED) use among adult patients seen at Geisinger's Community Medicine Service Line (CMSL) clinics. The intervention occurs immediately following an appointment where a patient receives a diagnosis of an ambulatory sensitive condition (ASC; i.e., a condition considered to be a risk factor for near-term ED use). The evaluation will compare eligible patients with an ASC who were randomly assigned to receive follow-up outreach from a nurse (who was automatically prompted via the Epic electronic health record system to initiate outreach) with those who were randomly assigned to receive standard care. Analyses will be intent-to-treat. The primary outcome is ED use in the week following the appointment.

#### **Objectives**

The study will evaluate an intervention aimed at reducing ED use following ASC diagnoses via nurse post-appointment calls. Analyses will assess whether ED use is lower in the patients receiving the intervention vs. those in the control arm.

#### Design

This study is a randomized controlled trial with two study arms. Patients will be randomized to have their nurses receive or not receive outreach via Epic (the night following their appointment).

#### **Methods**

At the end of an eligible patient's CMSL appointment, a patient will be assigned to one of the following study arms, based on which of several ranges of randomized numbers that patient was originally assigned in their electronic chart:

**Current standard practice (control arm):** Patients will not be included in a nurse follow-up call list.

**Nurse nudge:** Following their visit and ASC diagnosis, patients in this arm will be included on an automated list for a nurse follow-up call. Note that, although the nurses will be prompted to call, not all patients in this arm will receive a call.

#### **Power Analysis**

With 2,988 patients, we would have 80% power to detect a 1.2% absolute decrease in ED visits between the active arm and the control arm, with two-tailed alpha of .05, assuming a 2% baseline rate of subsequent ED visits within 7 days. The target effect size and baseline rate were taken from a similar intervention on a separate service line at Geisinger.

#### **Project Status**

The intervention began on 1/6/2025. No data have been extracted from the electronic health record.

## **Statistical Analysis Plan**

### Planned Analyses

**Primary Outcome:** ED visit [Time Frame: within 7 days post-appointment]

Question: Does outreach decrease ED visits?

Analysis (Confirmatory): We will test the hypothesis that automatic Epic notification decreases the likelihood patients will visit the ED in the 7 days following the day of their appointment. We will run an OLS regression including a categorical predictor variable coding for experimental arm (0 = control arm, 1 = outreach arm).

**Other pre-specified outcome:** Nurse call to patient [Time frame: within 7 days post-appointment]

**Question:** Does the nurse nudge increase post-appointment nurse calls to patients?

Analysis (Confirmatory): We will test the hypothesis that automatic Epic notification increases the likelihood that nurses will call patients in the 7 days following the day of their appointment. We will run an OLS regression including a categorical predictor variable coding for experimental arm (0 = control arm, 1 = outreach arm).

#### **Analysis Notes**

Recent work suggests that OLS regressions are appropriate in randomized experiments with binary outcome variables such as ours (Gomila, 2021).

#### Reference

Gomila, R. (2021). Logistic or linear? Estimating causal effects of experimental treatments on binary outcomes using regression analysis. *Journal of Experimental Psychology: General*, 150(4), 700-709. https://doi.org/10.1037/xge0000920